CLINICAL TRIAL: NCT02835820
Title: The Effect of a Ketogenic Diet on HIV-Associated Neurocognitive Impairment
Brief Title: Effects of Diet on Brain Processing
Acronym: EDBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Shannon Morrison, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV and Diet Study
Record Dates: First submitted 2016-05-06; First posted 2016-07-18 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: HIV; Neurocognitive Impairment
Keywords: HIV; Neurocognitive; Ketogenic Diet
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketogenic Diet Group (Experimental): Ketogenic meals (3 meals/day, 7 days/week x 12 weeks) prepared and delivered to participants.
  Interventions: Dietary Supplement: Ketogenic Diet
- Patient Choice Diet (No Intervention): Control.

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — 12 week delivery of all meals/snacks (eucaloric) prepared by a registered dietician.
  Arms: Ketogenic Diet Group

SUMMARY:
Randomized control pilot 12 week feeding trial to compare the preliminary effects of ketogenic diet (versus patient choice diet) on HIV-associated neurocognitive impairment. N = 20 (n = 10/10) randomized to diet condition. Pilot data necessary to evaluate the feasibility and determine initial data for primary outcomes in order to accurately determine needed sample size for larger clinical trial.

Outcomes: 1) cognition (NIH Toolkit), 2) cardiometabolic markers (insulin glucose, insulin resistance, markers of inflammation), and 3) neural activity (as determined by functional MRI..

DETAILED DESCRIPTION:
Specific Aims: In medically stable, older (> 50 years) HIV patients with cognitive impairment, this study will:

Overall: Test the feasibility of recruitment, retention, and adherence to a ketogenic diet versus patient choice diet (PCD) intervention.

Primary: Compare the impact of a 12-week KD versus PCD on:

1. Cognitive function (at 12 weeks).
2. Inflammation (at 12 weeks).
3. Cardiometabolic profile (at 12 weeks).
4. Persistence of cognitive effects (at 18 weeks).

   Secondary: In a subsample (n = 5; experimental group):
5. Examine the changes in neural activity and neurocognitive functioning as demonstrated via magnetic resonance imaging (MRI), after a 12 week KD diet.
6. Assess the level of agreement between NIH Neurocognitive Tests and MRI in the assessment of neurocognitive functioning.

INNOVATION: Brain metabolism regulation and reduced neural inflammation via dietary approaches have only recently been explored in the treatment/management of progressive cognitive disorders in humans. Preliminary results in Alzheimer's and Parkinson's patients suggest that the use of ketones for brain fuel improves brain metabolism and cerebral perfusion as well as reduces accumulation of harmful brain proteins20 To date, the effects of a KD in cognitively impaired older HIV patients have not been explored. In addition, this study proposes the use of MRI testing to examine the longitudinal, physiologic changes in the brain of cognitively impaired, older HIV patients consuming a KD for 12 weeks. Moreover, this study will utilize the new FDA-approved Magnetom Prisma 3T MRI system to better visualize small-scale neural brain abnormalities.

Research Design and Methods Design/Setting: Using an experimental design, a total of 20 older (> 50 years), stable HIV participants (CD4+ lymphocyte count > 350 cells/mm3 for at least two years and prescribed their current cART regimen for at least six months) with self-identified "forgetfulness" and demonstrate cognitive impairment (score </= on Telephone Interview for Cognitive Status -Modified (TICS-M)) will be recruited from the 1917 clinic (data extracted/verified using 1917 Clinic database) and will be randomly assigned to either the ketogenic diet (KD)(< CHO 50 grams/day) (n = 10) or the patient choice diet (PCD) (no dietary restrictions/changes) (n = 10) group for 12 weeks. In addition, the first five (n = 5) eligible (i.e., no metal implants, claustrophobia) participants randomized to the experimental group will also be enrolled in an additional magnetic resonance imaging (MRI) longitudinal study to generate preliminary data regarding the neurological changes associated with cognitive improvement. Previous studies in Alzheimer's and Parkinson's disease patients have reported significant cognitive improvement at 28, 45, and 90 days of ketosis.

Exclusion Criteria: Current drug or alcohol abuse (> 3 drinks/day), past medical history of mental disorders (i.e., schizophrenia, bipolar), neural injury (i.e., cerebral vascular accident or traumatic brain injury), dementia, Parkinson's, diabetes mellitus, hearing impaired, or any other condition that contraindicates participation. Due to the inconclusive evidence regarding the influence of statin drugs on cognition, statin use will not be exclusionary.

Recruitment: Fliers that provide basic study and PI contact information will be posted in the lobby/exam rooms of the 1917 Clinic. A telephone screening interview will be completed for all interested individuals. During the screening, cognitive impairment will be determined via administration of the Telephone Interview for Cognitive Assessment-Modified (TICS-M). TICS-M is a 13-item tool for assessment of cognitive function in older adults. A score < 20 indicates cognitive impairment (equivalent to a score < 25 on the validated/widely used in-person cognitive assessment, Mini Mental Status Exam [MMSE]).

Randomization: Participants will be randomly assigned, using permutated block randomization, to either the KD or PCD group with equal size. The CCTS BERD methodologists will develop the permuted block randomization algorithm. Because this is a diet intervention, it is not possible for participants/study personnel to be blinded to group assignment. In order to minimize bias/ensure allocation concealment, the randomization schedule will include sequentially-numbered, opaque sealed envelopes and will be kept by Dr. Morrison.

Data Collection:

Demographics: Age, education, gender, marital/partner status, employment status/disability eligibility, SES (Medicaid, food stamps, p Public housing eligibility), years since HIV diagnosis (baseline assessment only).

Anthropometrics: Height, weight, BMI, waist and hip circumference assessed at baseline and week 1. Height (nearest 0.1 cm), waist circumference (nearest 0.1 cm), and hip circumference (nearest 0.1 cm) measured with Gulick tape measure. Weight (nearest .01 kg) assessed using a Tanita body composition analyzer BC418, Tanita Corp of America, Arlington Heights, IL. BMI will be calculated. Waist circumference will be measured at the umbilicus at end of inspiration. Hip measures will be evaluated at widest hip portion.

Cognition: Cognition will be determined via the well-validated NIH Cognition Toolbox Battery. The NIH Toolbox is a comprehensive computerized battery that assesses each major cognitive domain in ~30 minutes. This technology has been in design/beta testing for nearly a decade by world-renowned neuropsychologists and computer programmers. Scoring includes the following corrected (age, education, gender, race) scores: fluid cognition composite, crystalized cognition composite, overall cognitive function composite, and scores for each individual domain (i.e., executive function, attention, episodic memory, language, processing speed, and working memory). Impairment scores can be derived from each of the aforementioned scores.

Neuroimaging: All neuroimaging screening, data collection, and data analyses will be conducted by Dr. Jarred Younger. Approved participants will attend a baseline imaging session. All imaging will be performed on the UAB Civitan International Research Center's 3-Telsa Siemens Prisma scanner and 64-channel head/neck receiving coil. Participants will first complete a high-resolution structural scan for group registration. Participants will then complete the T2*-weighted blood oxygen level dependent (BOLD) functional scan. The functional scan will use a "resting-state" protocol in which the participants are instructed to close their eyes and rest. The 12-minute run will collect functional volumes every 2 seconds. Participants will be invited back to the scanner after completing the intervention, at which time they will repeat the entire scan sequence. Structural and functional data will be examined longitudinally to determine changes occurring as a result of the intervention. Changes in gray-matter structure will be examined using a high-dimensional warping (HDW) tensor-based morphometry approach. Functional data will be analyzed using a Fractional Amplitude of Low Frequency Fluctuations (FALFF) approach. The relative activity pattern will be contrasted in the pre-intervention and post-intervention scans to determine areas showing greater or lesser neural activity after the intervention diet. To help mitigate the loss of statistical power due to the low sample size in this preliminary analysis, all statistics will be run within-person with a voxel-wise statistical threshold of p < 0.005.

Oral Glucose Tolerance Test (OGTT): Screening consists of a glucose load of 75 g at baseline (time 0). At ~7 am, after a 12-h fast, a flexible intravenous catheter will be placed in an antecubital space. Blood samples will be collected at times 0, 10, 20, 30, 60, 90, and 120 minutes. Sera will be stored at -85oC until analyzed for glucose, insulin, and C-Peptide. Whole-body insulin sensitivity and β cell responsiveness will be derived via OGTT at baseline/week 12.

Analysis of Glucose, C-peptide, and Insulin: Concentrations of glucose, insulin, and C-peptide will be analyzed in the UAB Diabetes Research Center (Core Director: B. Gower, Primary Mentor). Glucose will be measured in 3 µL sera using the Glucose oxidase method on a Stanbio Sirrus analyzer (Stanbio Laboratory, Boerne, TX). Insulin will be assayed in 50-µL aliquots using immunofluorescence on a TOSOH AIA-II analyzer (TOSOH Corp, S. San Francisco, CA). C-peptide will be assayed in 20-µL aliquots using the TOSOH analyzer.

Lipids: Total, high density cholesterol (HDL) and triglycerides will be measured using SIRRUS analyzer (Stanbio Laboratory, Boerne, TX); low density lipoprotein will be calculated using the method of Friedewald.

Inflammation Markers: Assessed by immunoassay in fasting morning sera before and after the intervention. High-sensitivity C-reactive protein (CRP) will be assessed by turbidometric methods by using a SIRRUS analyzer (Stanbio Laboratory), with reagents obtained from Pointe Scientific, and TNF-a and IFNy, IL-1B, IL-6, IL-8, and IL-12p70 by using electrochemiluminescence (Meso Scale Discovery).

Urine Ketones: Presence of acetoacetic acid (ketones) assessed via Precision XTRA Ketone Monitoring System. All participants will monitor capillary glucose daily for first two weeks and then weekly. Results will be documented on log sheet and returned to study staff. Participants will be contacted via telephone on weeks 4 and 8 to remind of ketone log submission.

Procedures: Eligible participants will be randomized to either the experimental (n = 10) or control group (n = 10) and scheduled for baseline data collection. Laboratory, demographic, and anthropometric assessments will be completed UAB's Clinical Research Unit (CRU). Baseline data will include: demographic questionnaire, oral glucose tolerance test (OGTT), inflammatory assays and lipid panel as well as an anthropometric evaluation. In addition, participants will be provided training related to the assessment of urine ketones, including a visual aid/handout that displays the color rubric and corresponding numeric value. Even though all snacks and meals for the KD group will be provided, experimental group participants will receive nutritional counseling related to the KD and provided with handouts that highlight important components of a KD so that participants can remain adherent to the intervention even if eating in a restaurant or in other social settings. After completion of the aforementioned items, participants will be escorted to the UAB Hospital cafeteria and provided a voucher for breakfast prior to completion of cognition assessments. After breakfast completion, participants will return to the CRU for completion of the cognitive battery in a private conference room. Completion of the questionnaires will be completed on a laptop computer that is secured by PGP Whole Disk Encryption® software to ensure participant confidentiality/privacy. After completion of the cognitive battery, individuals randomized to the experimental group and willing/eligible to undergo MRI testing, will be escorted to the UAB Highlands radiology department. Delivery of meals/snacks (week 1) will begin the week following baseline data collection. Bi-weekly phone conferences will be conducted with all participants to maintain participant contact as well as to assess for intervention adherence, challenges, and answer questions. In addition, all participants will complete a urine ketone assessment on weeks 4 and 8 and report those findings during conference calls. Note: Participants prescribed medications known to cause abnormal urine color (i.e., azo dyes, nitrofurantoin, and riboflavin) or affect the results (levodopa, hydroxyquinoline , methyldopa/captopril) or who report difficulty distinguishing differences between colors will return to UAB's CRU for serum ketone analysis at weeks 4 and 8. In addition, a survey will be administered to the KD group to determine what participants liked and did not like about the diet (week 12). All participants will be compensated for their time as follows: 1) Baseline and post intervention (wk 12) laboratory and cognitive assessments, $50/visit (N = 20); 2) MRI completion (n = 5), $50/scan; 3) Ketone assessment (wks 4 and 8, n = 20), $10 each; and 4) Six-week post intervention cognitive assessment (wk 18), (N = 20), $25.

Dietary Intervention:

KD: Meals/snacks will be provided/prepared by the UAB Clinical Research Unit's Bionutrition Department, a unit that employs two Dietitians who are all registered through the Academy of Nutrition and Dietetics and licensed in their perspective states. Food will be delivered weekly via a courier in appropriate food transportation coolers. The UAB Bionutrition Department is has a wealth of experience in research feeding study implementation including studies requiring specialized meal plans. Meals will be matched for energy content to maintain current energy balance and consist of < 50 grams CHO/day. Daily CHO intake will primarily be derived from fresh vegetables.

PCD group: Participants in this group will be instructed to maintain their normal dietary patterns. To ensure control group participants are not electively consuming a ketogenic diet (< 50 g CHO/day) during the 12 week intervention, participants will complete an at-home urine ketone screen and report results to project coordinator or PI on weeks 4 and 8. If a ketogenic diet is electively being consumed by a member of PCD group, the participant will be allowed to complete the study; however, the participant's data won't be included in analyses.

Intervention Fidelity: Intervention fidelity will be assessed using strategies consistent across the literature. 31-34 35 A comprehensive manual will be developed detailing recruitment, retention, assessment, and standardized intervention protocols. Standardized checklists will be utilized to review procedures. When a checklist item is not met, reasons will be explored/re-training will occur. Each participant will be contacted by telephone biweekly to reinforce intervention concepts (based on group assignment), appointment reminders, answer questions, and address areas of concern. Intervention adherence will be assessed at weeks 4 and 8 via urine ketone analysis unless contraindicated which, in case, serum ketones will be analyzed.

Statistical Analysis:

Demographic, Anthropometrics and Baseline Characteristics: Demographic data (i.e., age, education, gender, marital/partner status, employment status, and years since HIV diagnosis; anthropometrics (i.e., height, weight, BMI, waist and hip circumference); and baseline measures including cognition (cognitive scores and impairment score), inflammatory markers (CRP, TNF-a, IFNy, IL-1B, IL-6, IL-8, and IL-12p70), cardiometabolic factors (OGTT, glucose, C-peptide, and insulin) will be reported for each subject. Comparisons between the diet groups will be conducted to assess the degree to which comparability of randomization was achieved.

Primary analysis: All the primary outcomes (impairment score, inflammatory markers and cardiometabolic factors) will be examined by an analysis of covariance (ANCOVA) including the change from baseline to completion of diet treatment as dependent variable, study group as independent variable, and baseline measures as a covariate, to evaluate the effects of a 12 week KD versus PCD. The lasting cognitive effects of a 12 week KD versus PCD six weeks post intervention completion will be examine by an ANCOVA including the change of impairment score form 12 week to 18 week as dependent variable, study group as independent variable, and impairment score at 12 week as a covariate.

Secondary analysis: The changes in neural activity and neurocognitive functioning as demonstrated via MRI in the subsample of KD group will be examined by a paired t test. Spearman R correlation will be conducted to assess level of agreement between NIH Neurocognitive Tests and MRI in the assessment of neurocognitive function in medically stable HIV patients aged > 50 years.

Next steps: An important reason for conducting this pilot study is to evaluate the feasibility and determine initial data for the primary outcomes, in order to perform a sample size calculation for a larger trial. The mean and the standard error of the difference between the changes of KD group and PCD group will be used for the sample size calculation to reach an 80% power. In addition, the study protocol, data collection questionnaires, randomization procedure, recruitment and consent, and acceptability of intervention will be evaluated. Findings and the tested/improved protocol of this study will support an R21/R01 mechanism (i.e., PAR-15-280/PAR-15-282: Multidisciplinary Studies of HIV and Aging) that will include and expand upon following specific aim and hypotheses:

Specific aim: Compare the cognitive, cardiometabolic, and neural structural effects of a KD versus PCD in medically stable, older (> 50 years) HIV patients with cognitive impairment.

It is postulated that, in comparison to the control group, older (aged > 50 years) HIV positive, cognitively impaired individuals randomized to the KD will demonstrate the following:

Hypothesis 1: Improved cognition. Hypothesis 2: Decreased insulin, glucose, and systemic inflammation as well as improved insulin sensitivity.

Hypothesis 3: Heightened neural activity as observed by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Stable HIV participants (CD4+ lymphocyte count > 350 cells/mm3) for at least two years
* prescribed their current cART regimen for at least six months) with mild to moderate cognitive impairment

Exclusion Criteria:

* Drug/alcohol abuse
* History of Parkinsons
* Alzheimers, stroke or traumatic brain injury
* diabetes mellitus
* renal insufficiency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Morrison, PhD, Principal Investigator — Faculty
Locations (1):
- UAB 1917 Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Morrison SA, Fazeli PL, Gower B, Willig AL, Younger J, Sneed NM, Vance DE. Cognitive Effects of a Ketogenic Diet on Neurocognitive Impairment in Adults Aging With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2020 May-Jun;31(3):312-324. doi: 10.1097/JNC.0000000000000110. PMID 31725105

RESULTS

PARTICIPANT FLOW:
Groups:
- Participant Choice Diet: Control. Participants maintained normal dietary behaviors
Period: Overall Study
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Started | 7 | 10
Baseline Screen (OGTT) | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 3
Not completed — Baseline Screen Failure | 0 | 3

BASELINE CHARACTERISTICS:
Population: Three participants dropped out of the patient choice diet due to baseline screen failure.
Groups:
- Patient Choice Diet: Consumes regular diet/no diet restrictions
- Total: Total of all reporting groups
Arm/Group | Ketogenic Diet Group | Patient Choice Diet | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (5.7) | 54.3 (4.7) | 55.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Food Insecurity [Count of Participants; unit: Participants] | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Neurocognition: Mean Score of Hopkins Verbal Learning Test (Total) at Baseline
Description: The Hopkins Verbal Learning Test is used to measure episodic verbal learning and memory. The range of the score for the Hopkins Verbal Learning score is as follows: > 130 superior; 120-129 high; 110-119 bright, normal; 90-109 average; 85-89 low average; 70-84 borderline mental deficit; 35-49 moderate mental deficit; 20-34 severe mental deficit; 20-25 profound mental deficit.
Time Frame: baseline
Population: Three participants from the PCD ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 29.4 (9.8) | 31.1 (8.6)

2. Primary Outcome: Neurocognition: Mean Score of Hopkins Verbal Learning Test (Total) at 12 Weeks Post Baseline
Description: as for outcome 1
Time Frame: baseline to week 12
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 35.3 (9.6) | 34.9 (12.6)

3. Primary Outcome: Neurocognition: Mean Score of Hopkins Verbal Learning Test at 18 Weeks Post Baseline
Description: as for outcome 1
Time Frame: baseline to week 18
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 39.6 (9.1) | 36.6 (11.7)

4. Primary Outcome: Neurocognition: Mean Score of Wechsler Adult Intelligence Scale at Baseline
Description: The Wechsler Adult Intelligence Scale is an II test to measure intelligence and cognitive ability. The Full Scale scores are: beyond 130 place an individual in the superior or gifted range; scores between 120-129 suggest very bright; scores between 110-119 are bright normal; scores as 90-109 are average; scores of 85-89 suggest average intelligence; score of 70-84 suggests low average intelligence; score of 50 - 69 suggests borderline mental functioning; score of 50 - 69 suggests mild mental retardation; score of 35-49 suggests moderate retardation; 20 - 34 suggests severe retardation; below 20 - 25 suggests profound retardation
Time Frame: baseline
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 46.1 (9.3) | 46.0 (7.5)

5. Primary Outcome: Neurocognition: Mean Score of Wechsler Adult Intelligence Scale at 12 Weeks Post Baseline
Description: The Wechsler Adult Intelligence Scale is an I! test to measure intelligence and cognitive ability. The Full Scale scores are: beyond 130 place an individual in the superior or gifted range; scores between 120-129 suggest very bright; scores between 110-119 are bright normal; scores as 90-109 are average; scores of 85-89 suggest average intelligence; score of 70-84 suggests low average intelligence; score of 50 - 69 suggests borderline mental functioning; score of 50 - 69 suggests mild mental retardation; score of 35-49 suggests moderate retardation; 20 - 34 suggests severe retardation; below 20 - 25 suggests profound retardation
Time Frame: baseline to 12 weeks
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 46.7 (8.1) | 46.1 (9.5)

6. Primary Outcome: Neurocognition: Mean Score of Wechsler Adult Intelligence Scale at 18 Weeks Post Baseline
Description: as for outcome 5
Time Frame: baseline to 18 weeks
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 52.0 (10.8) | 44.7 (10.2)

7. Primary Outcome: Neurocognition: Mean Score of Trail Making A and B at Baseline
Description: Trails A (simple) and Trails B (alternative) neuropsychological assessments provide information on cognitive processes such as visual search, scanning, speed of processing, mental flexibility, and executive functions (i.e., memory, problem solving, verbal reasoning). It is sensitive to cognitive impairment associated with dementia. The average score for trail making is 29 seconds. Scores over 78 seconds suggest a deficit.
Time Frame: baseline
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: Seconds to complete
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
Seconds to complete | 41.6 (17.0) | 50.0 (7.7)

8. Primary Outcome: Neurocognition: Mean Score of Trail Making A and B at 12 Weeks Post Baseline
Description: Trails A (simple) and Trails B (alternative) neuropsychological assessments provide information on cognitive processes such as visual search, scanning, speed of processing, mental flexibility, and executive functions (i.e., memory, problem solving, verbal reasoning).It is sensitive to cognitive impairment associated with dementia. The average score for trail making is 29 seconds. Scores over 78 seconds suggest a deficit.
Time Frame: baseline to 12 weeks
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: Seconds to complete
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
Seconds to complete | 44.6 (17.6) | 44.3 (8.3)

9. Primary Outcome: Neurocognition: Mean Score of Trail Making A and B at 18 Weeks Post Baseline
Description: as for outcome 7
Time Frame: baseline to 18 weeks
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: Seconds to complete
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
Seconds to complete | 40.1 (16.2) | 44.1 (11.9)

10. Primary Outcome: Neurocognition: Mean Score of Stroop Test at Baseline
Description: The score of greater than is considered normal; a score of 40 or less is considered "low" whereas a score greater than 40 is considered "normal".
  Stroop test is named after the instrument developer, John Stroop. The instrument title is not an acronym.
Time Frame: baseline
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: Number of correctly identified items
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
Number of correctly identified items | 36.3 (6.8) | 36.0 (6.0)

11. Primary Outcome: Neurocognition: Mean Score of Stroop Test at 12 Weeks Post Baseline
Description: as for outcome 10
Time Frame: Baseline to 12 weeks
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: Number of correctly identified items
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
Number of correctly identified items | 40.0 (8.6) | 39.4 (6.2)

12. Primary Outcome: Neurocognition: Mean Score of Stroop Test at 18 Weeks Post Baseline
Description: The STROOP measures brain damage. The score of greater than is considered normal; a score of 40 or less is considered "low" whereas a score greater than 40 is considered "normal".
  Stroop test is named after the instrument developer, John Stroop. The instrument title is not an acronym.
Time Frame: baseline to 18 weeks
Population: Three PCD participants ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: Number of correctly identified items
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
Number of correctly identified items | 39.1 (8.1) | 40.1 (6.3)

13. Primary Outcome: Cardiometabolic Markers: Mean Fasting Glucose Measures at Baseline
Description: A fasting blood sugar level less than 100mg/dl is normal. A fasting blood sugar level of 100- 126mg/dl is considered prediabetic. 126mg/dl or greater suggests diabetes
Time Frame: baseline
Population: Three PCD participants were ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
mg/dL | 97.0 (1.4) | 101.4 (11.5)

14. Primary Outcome: Cardiometabolic Markers: Mean Fasting Glucose Measures at 12 Weeks Post Baseline
Description: as for outcome 13
Time Frame: baseline to 12 weeks
Population: Three PCD participants were ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
mg/dL | 98.1 (6.3) | 100.6 (16.6)

15. Primary Outcome: Cardiometabolic Markers: Mean Markers of Inflammation (C-reactive Protein) Measures at Baseline
Description: C-reactive protein (CRP) , a protein in the blood, indicates inflammation, specifically in the heart.. CRP levels rise with inflammation. A CRP concentration of below 1.0 mg/L indicates low risk; 1.0 to 3.0 mg/L suggests an average risk. Greater than 3.0 mg/L suggests a high risk.
Time Frame: baseline
Population: Three PCD participants were ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
mg/L | 11.33 (15.9) | 4.1 (1.9)

16. Primary Outcome: Cardiometabolic Markers: Mean Markers of Inflammation (C-reactive Protein) Measures at 12 Weeks Post Baseline
Description: as for outcome 15
Time Frame: baseline to 12 weeks
Population: Three PCD participants were ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
mg/L | 9.1 (10.2) | 3.6 (3.5)

17. Primary Outcome: Tumor Necrosis Factor Alpha (TNF or TNF-α)
Description: Tumor Necrosis Factor Alpha (TNF or TNF-α) is a major pro-inflammatory cytokine involved in inflammatory events. Being one of the most important pro-inflammatory cytokines, TNF-α participates in vasodilatation and edema formation, and leukocyte adhesion to epithelium through expression of adhesion molecules; it regulates blood coagulation, and also contributes to oxidative stress in sites of inflammation.
Time Frame: baseline
Population: Three PCD participants were ineligible due to baseline screen fail.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
pg/mL | 2.9 (1.3) | 3.0 (1.3)

18. Primary Outcome: Tumor Necrosis Factor (TNF or TNF-α)
Description: as for outcome 17
Time Frame: baseline to week 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 7 | 7
pg/mL | 2.7 (1.1) | 3.0 (0.9)

19. Secondary Outcome: Neural Activity: Presence or Absence of Impaired Bloodflow in the Brain at Baseline as Determined by a Functional MRI
Description: Functional MRI is used to determine blood flow in the brain. Absence of blood flow impairment will be recorded as '0' and impairment will be recorded as '1'
Time Frame: baseline
Population: Those randomized to intervention group at baseline without MRI contraindications
Measure: Count of Participants; unit: Participants
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

20. Secondary Outcome: Neural Activity: Presence or Absence of Impaired Bloodflow in the Brain at 12 Weeks Post Baseline as Determined by a Functional MRI
Description: as for outcome 19
Time Frame: Baseline to 12 weeks
Population: Intervention group as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
Number analyzed (Participants) | 3 | 0
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected across the 18 week study.
Description: One participant was admitted to hospital for asthma exacerbation.
Arm/Group | Ketogenic Diet Group | Participant Choice Diet
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketogenic Diet Group (N=7) | Participant Choice Diet (N=7)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient was admitted due to asthma exacerbation for 23-hour observation.

LIMITATIONS AND CAVEATS:
Small sample size (pilot study), limited ability to monitor intervention fidelity, no reassessment until 12 weeks thus it is unclear as to when cognitive benefits emerged in persons randomized to the KD group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT02835820/Prot_SAP_ICF_000.pdf